CLINICAL TRIAL: NCT00374569
Title: Dynamic Posturographic Testing and Motor Learning Predictability in Gymnasts
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal Investigator, Carrick Institute for Graduate Studies
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CI-05-05
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Gymnastics Injury, Motor Learning, Balance
Keywords: Gymnastics, Computerized Dynamic Posturography, Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gymnastics (Experimental): Gymnasts stand on a computerized dynamic posturography Force Plate and Stability is measured and gymnastic routines performed
  Interventions: Procedure: Gymnastic Routine
- Non Gymnasts (Experimental): Non Gymnasts stand on a computerized dynamic posturography Force Plate and Stability is measured and gymnastic routines performed
  Interventions: Procedure: Gymnastic Routine

INTERVENTIONS:
Procedure: Gymnastic Routine — A combination of gymnastic movements are performed

SUMMARY:
One aim of this study was to find if there was a difference between balance and stability between elite level gymnasts and non-gymnasts. Another aim was to find if there was a relationship between dynamic posturographic scores associated with sway fatigue or adaptability and the ability to learn new gymnastic routines. The ultimate aim of the study was to improve gymnastic performance while reducing the probability of injury.

DETAILED DESCRIPTION:
Computerized dynamic posturography outcomes will be obtained on elite level gymnasts and non gymnasts who will be age matched. The outcome measurement will be obtained using computerized dynamic posturography, a standard diagnostic test of balance function (41-46). The subject's balance was tested using a three-component force platform (CAPS test) under one sensory condition of the modified Clinical Test of Sensory Interaction on Balance (mCTSIB), the eyes closed on perturbing surface condition. This condition was chosen as studies have shown it to be the single test that best correlates with balance impairment and falls. The stability score, already used in several studies by other authors will be used as the primary outcome measure in this research. It is defined as 1 minus the ratio between the measured sway during the test (computed as the major axis of a standard 95% confidence ellipse) and the amount of sway a normal subject of the same height as the one being tested should be able to sway before falling (also known as the theoretical maximum sway or the theoretical limit of stability, calculated using a regression formula based on the subject's height developed by NASA in 1962 and commonly used in all posturographic tests). For convenience, the stability score will be expressed as a percentage. Its definition makes it a convenient and easy to understand measure to use as a subject able to stand perfectly still with no sway will have a score of 100%, whereas one that sways as much as the limit of stability will have a score of 0%. During each test, the subject's sway will be determined by the force platform and its related software. The CAPS three-component force platform uses 3 load cells arranged in a triangle to measure the distribution of the vertical ground reaction force on the platform. The analog load cell signals are amplified and simultaneously sampled by the platform electronics using three synchronized individual 24bit delta-sigma analog to digital converters sampling at 312kHz and decimating the samples to a data rate of 64Hz. The use of three A/D converters insures that the signals from the 3 load cells are acquired simultaneously with no timing error. The high sampling rate with the high decimation and low data rate of the sigma-delta converters eliminates aliasing and provides a resolution of about 4 parts per million. The digital load cell data was then sent via a USB connection to the PC where software uses a calibration matrix determined by the manufacturer to compute the total vertical force and the two horizontal moments acting on the platform. From these data, the software computed the point of application of the vertical force acting on the platform, commonly referred to as the Center of Pressure (CoP). The location of the CoP coincides in static conditions with the projection of the subject's Center of Mass (CoM) onto the platform, and its movement relates to the movements of the subject's CoM (sway). The determination of the actual sway will require the determination of the instantaneous location of the CoM via the location and inertial properties of each body segment of the specific subject being tested. The CAPS test, like all posturographic equipment, uses the movement of the CoP as an approximation of the sway. Because it is an approximation, and because for kinetic reasons the CoP moves more than the CoM, the 95% confidence interval of the CoP motion was considered. This will allow the CAPS software to compute the ellipse that represents the location of all of the sway samples collected during the test with 95% confidence. The major axis of this ellipse will represent the maximum sway of the subject in any direction during the test and it will be used to compute the stability score. To assess the accuracy and resolution of the measurement chain, calibrated weights of 75kg and 100kg will be positioned in the center of the force platform (as if it were a subject) and 20s acquisitions will be performed: the accuracy of the weight must be within the instrument's factory specifications (+-2N). Therefore the accuracy for the position claimed by the manufacturer of +-1mm for a weight of 75kg will be accepted as correct as it determination will require specialized equipment and software available only to the manufacturer. It should be noted that the overall accuracy of the position of the CoP given by the instrument will not be relevant in this study as the motion of the CoP determined the sway. The sway measurement error will be estimated considering the fact that during the test at both weights the dead weight must not move, but the measurement chain will indicate a "sway" of less then 0.05mm (measurement noise), therefore the resolution of the measurement chain and the sway measurement error will be considered to be 0.05mm. To verify the repeatability of the measurement chain, the same type of tests will be repeated two times, obtaining similar results (within the specified accuracy and resolution). Given the sway measurement error, the measurement error in the stability score will be determined. From the definition of the stability score it is clear that the least the theoretical limit of stability, the more pronounced the effect of the sway measurement error is. As the theoretical limit of stability is computed by using the formula 0.55*height*2*sin(6.25°), the shorter the subject, the more the stability score is sensitive to the measurement errors. To estimate the stability score measurement error a subject's height of 1.6m will be considered. Such a subject will have a theoretical limit of stability of 191.6mm. For such a subject, a sway measurement error of 0.05mm means a stability score measurement error of 0.05/191.6 or, if the score is expressed in percentage, of 0.026%. Thus, any changes in the stability score greater than that will be a consequence of the subject's sway and not of measurement errors. A CAPS dynamic posturography test in the eyes closed perturbed stance will be obtained on all subjects. Subjects will be instructed that they will stand on a foam platform and close their eyes while data will be obtained from a computerized force plate. The subjects will be given practice sessions so that they will be familiar with the test prior to the collection of data. The CAPS test occurs over 25 seconds. We will divide the degree of sway observed during the first half of the test and the second half of the test and will obtain ratios. Subjects whose sway will increase in the second half of the test in reference to the first half will be identified as demonstrating a fatigability ratio. Individuals who will demonstrate less sway in the second half of the test will be identified as demonstrating an adaptability ratio that we consider might be related to some type of motor learning. All gymnasts will be instructed in a novel gymnastic routine which will include a variety of inverted postures and ground routines unfamiliar to the subjects. The athletes will be allowed to practice the routine for one hour after which they will be asked to perform the routine in front of the same judge who will be blinded as to the outcome measures previously obtained. The performance scores will be then compared to the CDP measurements to ascertain if there would be any relationship.

ELIGIBILITY:
Inclusion Criteria:

* Elite level Gymnasts
* Non Gymasts control

Exclusion Criteria:

* Non Elite level Gymnasts

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2005-06; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Dynamic Posturography | pre and post
  stability testing pre and post gymnastic routines

SECONDARY OUTCOMES:
Blinded expert judging of motor performance in Gymnastics | pre and post immediate
  Judging of gymnastic performance

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, FACCN, Study Chair — Carrick Institute for Graduate Studies; Guido Pagnacco, PhD, Principal Investigator — Carrick Institute for Graduate Studies; Elena Oggero, PhD, Principal Investigator — Carrick Institute for Graduate Studies; Brandon Brock, DC, Study Chair — Carrick Institute for Graduate Studies; Tina Arikan, DC, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Carrick Institute for Graduate Studies Texas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrick FR, Oggero E, Pagnacco G, Brock JB, Arikan T. Posturographic testing and motor learning predictability in gymnasts. Disabil Rehabil. 2007 Dec 30;29(24):1881-9. doi: 10.1080/09638280601141335. Epub 2007 Feb 9. PMID 17852265